CLINICAL TRIAL: NCT00532324
Title: A Prospective Cohort Pilot Study of the Clinical and Molecular Epidemiology of Staphylococcus Aureus in Pregnant Women at the Time of Group B Streptococcal Screening in a Large Urban Medical Center in Chicago, IL USA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Thrasher Research Fund (Other); Northwestern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tina Q. Tan, Attending Physician, Division of Infectious Diseases, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2007-13145(CMH)/2623-001(NU)
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Staphylococcus Aureus
Keywords: Methicillin resistant Staphylococcus aureus; Staphylococcus aureus; Healthy term and near term neonates; Prevention; Nasal and Vaginal Colonization rates; Pregnant women
MeSH Terms: conditions — Staphylococcal Infections | interventions — Mupirocin; Triclosan; Sodium Hypochlorite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (No Intervention): Pregnant women not receiving CA-MRSA decolonization therapy.
- B (Other): Pregnant women receiving CA-MRSA decolonization therapy.
  Interventions: Other: CA-MRSA Decolonization

INTERVENTIONS:
Other: CA-MRSA Decolonization — In later stages of this study, women found to be nasally and/or vaginally colonized with CA-MRSA will be randomized to receive postpartum, either: 1) attempted decolonization with intranasal mupirocin twice a day for one to two weeks with or without diluted chlorhexidine or Clorox baths two to three times a week for one to two weeks or, 2) no intervention. The primary study is observational only.
  Other Names: Mupirocin also known as Bactroban; Chlorhexidine also known as Phisohex, Clorox
  Arms: B

SUMMARY:
Background:

Community acquired methicillin-resistant Staphylococcus aureus (CA-MRSA) is an emerging pathogen of the 21st century whose incidence as a cause of local and invasive infections has significantly increased, especially in previously healthy term and near term newborns. The etiology of the increasing incidence of infection in previously healthy term and near-term newborns remains unclear.

Hypothesis:

1. The incidence of previously healthy newborns infected with CA-MRSA skin & soft tissue (SSTI) and invasive infections is higher in those born to mothers colonized with CA-MRSA.
2. Pregnant women colonized with CA-MRSA are at higher risk for post-partum infection with this organism.

Specific Aims:

1. To determine the incidence of nasal and vaginal colonization with CA-MRSA in pregnant women and determine the genetic similarities of these strains.
2. To study CA-MRSA transmission dynamics and evaluate the incidence of SSTI and invasive infections in newborns born to S. aureus colonized mothers.
3. To study the efficacy of attempted decolonization in CA-MRSA colonized mothers in decreasing the incidence of transmission and development of SSTI and invasive infections in their infants during the first month of life.

Potential Impact:

Understanding the epidemiology of the transmission dynamics of CA-MRSA in previously healthy newborns will provide important information to support the development of strategies aimed at the interruption of transmission and prevention of infection caused by CA-MRSA in newborns, as well as in pregnant women. This will also allow for the development of infection control strategies to prevent the spread of this organism among post-partum units and nurseries.

DETAILED DESCRIPTION:
Background:

Community acquired methicillin-resistant Staphylococcus aureus (CA-MRSA) is an emerging pathogen of the 21st century whose incidence as a cause of local and invasive infections has significantly increased, especially in previously healthy term and near term neonates where it may be associated with high morbidity and mortality(1, 2, 3). The etiology for this increase remains unclear, but may be a consequence of perinatal or postnatal acquisition via maternal transmission through skin, breast milk, or vaginal colonization(4).

The major goals of our study are: to determine the incidence of pregnant women who are colonized with CA-MRSA, gain a better understanding of the transmission dynamics of this organism between the mother and the newborn infant, and to develop strategies for the prevention of transmission, spread and infection with this organism in both these populations.

This staged study is a collaborative effort between investigators from the Children's Memorial Hospital Division of Infectious Diseases, Northwestern Memorial Hospital Department of Obstetrics and Gynecology, and the Northwestern Memorial Hospital Division of Infectious Diseases. Collaboration across multiple specialties provides strength to the study by allowing the investigators to address multiple issues that are pertinent to both the care of pregnant mothers and newborn infants in the inpatient and outpatient setting.

Hypothesis:

1. The incidence of previously healthy term and near-term neonates infected with CA-MRSA skin & soft tissue (SSTI) and invasive infections is higher in those born to mothers vaginally and/or nasally colonized with CA-MRSA and, 2. Pregnant women vaginally and/or nasally colonized with CA-MRSA are at higher risk for post-partum infection with this organism.

Specific Aims:

1. To determine the incidence of nasal and vaginal colonization with CA-MRSA in pregnant women and determine the clonality of these strains.
2. To study CA-MRSA transmission dynamics and evaluate the incidence of SSTI and invasive infections in term and near-term newborns born to S. aureus vaginal and/or nasal colonized mothers.
3. To study the efficacy of attempted decolonization in CA-MRSA colonized mothers in decreasing the incidence of transmission and development of SSTI and invasive infections in their infants during the first month of life.

Methods:

1. Vaginal and anterior nasal cultures will be obtained prospectively over several months from pregnant women who obtain their prenatal care through Obstetrical practices at Prentice Women's Hospital and Maternity Center of Northwestern Memorial Hospital during the time of GBS screening at 34-36 weeks gestation. Together, these practices account for 300-500 deliveries per month.
2. Cultures will be plated on blood agar and incubated at 37oC for 48 hours. S. aureus strains will be identified by colony morphology and latex agglutination. MRSA isolates will be identified by PCR or latex agglutination for penicillin binding protein 2a by detecting the mecA gene and clonality by PFGE. PCR testing will then be used to identify strains carrying the Panton-Valentine Leukocidin gene as a marker of virulence.
3. In a prospective case-control cohort study, newborns born to CA-MRSA colonized mothers will have anterior nares cultures for S. aureus obtained at birth and followed for the development of SSTI and invasive infections for one month. Samples positive for MRSA will be tested for similarities to maternal isolates through methods described above. The newborn incidence of MRSA infection will be compared between those born to non-colonized mothers and those born to colonized mothers.
4. In further stages of this study, women found to be nasally and/or vaginally colonized with CA-MRSA will be randomized to receive postpartum, either: 1) attempted decolonization with intranasal mupirocin with or without diluted chlorhexidine or Clorox baths or, 2) no intervention.

Potential Impact:

Understanding the epidemiology of the transmission dynamics of CA-MRSA in previously healthy neonates will provide important information to support the development of strategies aimed at the interruption of transmission and prevention of infection caused by CA-MRSA in this patient population, as well as in pregnant women. This will also allow for the development of infection control strategies in the hospital setting to prevent the spread of this organism among post-partum units and nurseries.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women who present for routine OB/GYN care during the of the 34-36 week gestation GBS screening visit.
* Healthy term and near-term infants born to these mothers

Exclusion Criteria:

* Pre-term infants
* Infants who had significant illness after birth, i.e. transferred to neonatal intensive care unit for significant illness.

Age limits for infants will be 0-4 weeks of age and both genders will be included.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
CA-MRSA vaginal and nasal colonization rates in pregnant women at the time of routine Group B Streptococcus (GBS) Screening at 34-36 week gestation visit. | We will obtain vaginal and nasal samples at the 34-36 week gestation OB/Gyn visit.
The incidence of CA-MRSA skin, soft tissue and invasive (SSTI) infections in healthy term and near-term infants born to CA-MRSA colonized mothers. | Infants born to CA-MRSA colonized mothers will be followed for CA-MRSA colonization and/or SSTIs for the first 4 weeks of life.

SECONDARY OUTCOMES:
In later stages of the study, we will study the efficacy of attempted decolonization in CA-MRSA colonized mothers in decreasing the incidence of transmission and development of SSTI and invasive infections in their infants during the first month of life. | Infants born to CA-MRSA colonized moms will be followed for CA-MRSA colonization and/or SSTIs for the first 4 weeks of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Q Tan, M.D., Principal Investigator — Children's Memorial Hospital/Northwestern University Feinberg School of Medicine; Latania K Logan, M.D., Principal Investigator — Children's Memorial Hospital/Northwestern University Feinberg School of Medicine
Locations (1):
- Prentice Women's Hospital and Maternity Center of Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Kollef MH, Micek ST. Methicillin-resistant Staphylococcus aureus: a new community-acquired pathogen? Curr Opin Infect Dis. 2006 Apr;19(2):161-8. doi: 10.1097/01.qco.0000216627.13445.e2. PMID 16514341
- [Background] Crawford SE, Daum RS. Epidemic community-associated methicillin-resistant Staphylococcus aureus: modern times for an ancient pathogen. Pediatr Infect Dis J. 2005 May;24(5):459-60. doi: 10.1097/01.inf.0000164170.67897.97. No abstract available. PMID 15876949
- [Background] Deresinski S. Methicillin-resistant Staphylococcus aureus: an evolutionary, epidemiologic, and therapeutic odyssey. Clin Infect Dis. 2005 Feb 15;40(4):562-73. doi: 10.1086/427701. Epub 2005 Jan 24. PMID 15712079
- [Background] Fortunov RM, Hulten KG, Hammerman WA, Mason EO Jr, Kaplan SL. Community-acquired Staphylococcus aureus infections in term and near-term previously healthy neonates. Pediatrics. 2006 Sep;118(3):874-81. doi: 10.1542/peds.2006-0884. PMID 16950976